CLINICAL TRIAL: NCT04706624
Title: Screen, Treat and Retain Meth-using People With Opioid Use Disorders at Methadone Clinics
Acronym: STAR-OM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: University of California, Los Angeles (Other); University of Medicine and Pharmacy at Ho Chi Minh City (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Giang Le Minh, Associate Professor of Global Health; Deputy Director, Center for Training and Research on Substance Abuse-HIV (CREATA-H); Director, Office of Post-graduate Studies, Hanoi Medical University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HanoiMU; R01DA050486 (NIH)
Record Dates: First submitted 2021-01-04; First posted 2021-01-13 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Methamphetamine Abuse; Opioid-use Disorder; HIV Seropositivity
Keywords: methamphetamine use; opioid use disorders; methadone; HIV
MeSH Terms: conditions — Opioid-Related Disorders; HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: Two frontline interventions: contingency management (CM) throughout 12 weeks (high intensity CM); and CM in 6 weeks followed by 6 weeks of weekly group educational sessions (low intensity CM); Consecutive urine tests negative with methamphetamine at week 11 and week 12 (two urine tests per week) are considered as responsive to frontline interventions; any positive with one of the urine tests during week 11 and 12 or failure to provide urine are considered non-responsive; Three treatment alternatives: Responders to frontline interventions will receive two daily automatic unidirectional scripted SMS reminder plus one weekly self-monitoring assessment message over 12 weeks (maintenance treatment); non-responders will be randomized to either Matrix group counseling alone or Matrix group counseling with CM over 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity frontline intervention (Experimental): Participants who are assigned to the 12-week contingency management arm.
  Interventions: Behavioral: Contingency management (12 weeks); Behavioral: SMS reminders; Behavioral: Matrix only; Behavioral: Matrix + Contingency management
- Low intensity frontline intervention (Experimental): Participants who are assigned to the 6-week contingency management plus 6-week group education arm.
  Interventions: Behavioral: Contingency management (6 weeks); Behavioral: SMS reminders; Behavioral: Matrix only; Behavioral: Matrix + Contingency management; Behavioral: Group education (6 weeks)

INTERVENTIONS:
Behavioral: Contingency management (12 weeks) — Participants receive 12 weeks of contingency management.
  Arms: High intensity frontline intervention
Behavioral: Contingency management (6 weeks) — Participants receive 6 weeks of contingency management.
  Arms: Low intensity frontline intervention
Behavioral: SMS reminders — Participants receive two daily SMS reminders plus one weekly self-monitoring assessment.
Behavioral: Matrix only — Participants attend 12 weekly Matrix group counseling sessions.
Behavioral: Matrix + Contingency management — Participants attend 12 weekly Matrix group counseling sessions plus 12 weeks of contingency management.
Behavioral: Group education (6 weeks) — 6 weeks of group education
  Arms: Low intensity frontline intervention

SUMMARY:
The investigators propose to develop and evaluate optimal combinations of evidence-based interventions to improve HIV outcomes and reduce methamphetamine use (hereafter: meth use) among people with opioid use disorder who are in methadone maintenance therapy (MMT) in Vietnam. Over the past decade, the expansion of MMT has contributed to stemming both HIV and opioid epidemics. However, rising meth use threatens these achievements.

Evidence-based interventions such as Motivational Enhancement Therapy, Contingency Management, Matrix Model, and SMS reminders are effective in reducing meth use. The study will be conducted in the two largest cities in Vietnam, Hanoi and Ho Chi Minh City (HCMC), where there are the highest number of MMT patients and the highest burden of HIV cases. Building on the pilot work of the research team in Hanoi, through collaborative work with local MMT providers and patients, the investigators will first further refine adapted EBIs to develop adaptive strategies. The adaptive design includes: (1) Two frontline interventions: 6 weeks of contingency management then 6 weeks of weekly group educational sessions and 12 weeks of contingency management; (2) One (short-term) tailoring outcome: urine tests negative with meth metabolites in both week 11 and 12 are considered responsive to frontline interventions; (3) Three alternative interventions: those with positive outcomes will move to 12-week maintenance stage and receive two daily SMS reminders plus one weekly self-monitoring assessment messages. Non-responders will move to 12-week enhanced treatment stage and are randomly assigned to either Matrix group counseling only or Matrix group counseling plus contingency management.

The full randomization trial will be conducted with 200 HIV-positive and 400 HIV-negative MMT patients who report moderate- and high-risk meth use on self-screening with ASSIST or have urine positive with meth metabolites. In each location, the study will stratify participants by HIV status before randomizing them to one of two frontline interventions. Primary outcomes - including HIV viral suppression, HIV risk behaviors, and meth use (reported and urine tests) - will be assessed at 12, 24 and 48 weeks. The study team also conducts ethnographic observations and in-depth interviews with MMT clinic managers, clinical staff and MMT patients to explore implementation barriers and facilitators.

DETAILED DESCRIPTION:
1) To develop adaptive interventions, including two frontline interventions and four adaptive strategies, through collaborative processes (Aim 1): During Month 3 - 9, the investigators refine the EBIs to develop adaptive interventions.

1a) Assessment: The team conducts 4 Focus Group Discussions (FGDs) with MMT patients on local taxonomy and patterns of meth use, trigger situations, motivations for seeking treatment, motivations and barriers for participating in different EBIs, inputs/advice on proposed adaptive design, and barriers and facilitators for retention of participants in each of the adaptive steps.

1b) Decision: The team organizes a workgroup that involves MMT clinical staff, representatives of CBOs working with people who use drugs, social workers working with MMT patients, and MMT patients themselves to review the contents of FGDs in the Assessment step, experiences of pilot intervention in Hanoi, the conceptual and empirical evidence of EBIs to make recommendations on core contents of each EBI.

Contingency management is a 12-week or 6-week low-value escalating schedule. Participants give urine twice a week. Matrix group counseling involves twice weekly group sessions that last for about 60 to 90 minutes each. Group counseling focuses on relapse prevention. SMS-text: Participants receive automated, unidirectional, scripted, theory-based and culturally responsive text reminders twice daily plus a weekly self-monitoring assessment messages. The text messages are scripted across: 1) drug use, sexual risk reduction, physical health and HIV care (for HIV+ participants); and, 2) the theoretical construct of cognitive-behavioral therapy including understanding external and internal triggers; relapse prevention and relapse analysis and goal setting.

1c) Administration: At the end of the Decision step, the workgroup put together a framework for the adaptive design that include different interventions, sequence, decision rule and contents of interventions. This framework is presented and discussed in a second round of FGDs with target populations in each city.

2) Pilot implementation of adaptive interventions (Aim 1): During Month 3 - 9, the study team chooses one MMT clinic in each city for piloting the adaptive design. The pilot implementation, which lasts 12 weeks, aims to identify issues that need to be addressed before the full implementation. The pilot recruits 40 meth-using MMT patients (20 from each city, at least 10 HIV positive) and over-recruits women. Inclusion criteria for the pilot sample include: 1) 16 years old or older; 2) score of 4-26 (moderate risk) or 27+ (high risk) on ASSIST regarding meth use OR urine screen positive for metabolite of meth; 4) having a cell phone able to receive texts; (5) and willing to participate in treatment. These participants are excluded from the full implementation.

2a) Pilot Monitoring and Evaluation: The study team in each city monitors the overall operation of the pilot to ensure that interventions are carried out as planned. For each intervention session, a Master Behavioral Counselor and an ethnographer observe the implementation regarding content integrity, flow, location, message clarity, interventionist-participant interaction, participant attendance, engagement, and responsiveness. Second, after each phase of intervention implementation (self-screening, frontline interventions, decision stage, maintenance, enhanced treatment), a FGD is organized for all intervention facilitators and another with patients to understand their experiences and to gather feedback regarding potential modifications.

2b) Intervention modification and assessment finalization: The evaluation data helps to identify factors that may affect implementation and outcomes. Modifications to intervention characteristics to ensure the relevance of the intervention for target settings and populations are completed at this stage. This phase gives an opportunity to finalize the recruitment and retention strategies as well as assessment tools.

3) Full implementation of SMART design to compare effectiveness of two frontline interventions and four adaptive strategies (Aim 1) 3a) Selection of clinical settings to become intervention sites: Criteria for selecting clinics are established. Existing statistics are viewed and clinics that meet criteria are shortlisted. 20 MMT clinics are selected randomly from the shortlisted candidates (10 from Hanoi, 10 from HCMC).

3b) Intervention facilitator recruitment and training: The intervention team in each city includes one Master Behavioral Counselor with Master-level training in clinical psychology and two intervention coaches with bachelor degrees in social work, psychology or public health to support and ensure quality of implementation of the EBIs by MMT clinical staff. Both Master Counselor and intervention coaches are also facilitators for Matrix group counseling where MMT clinical staff will not be able to carry out themselves.

Once MMT clinics are selected, managers of these clinics nominate a physician, two counselors and one nurse to participate in the study as intervention facilitators. Before the start of intervention, all intervention staff at MMT clinics (1) receive didactic training on the theory behind the approach; (2) pass a knowledge test to evaluate their grasp of the concepts within and behind the approach; (3) watch a video of a Master Behavioral Counselor conducting intervention sessions and discuss the details of the session, and (4) conduct at least two pilot EBIs, which are recorded and observed by the HMU/UMP intervention team and the PIs. All subsequent interventions are audio recorded and coded to ensure the presence of essential elements of the intervention. Intervention staffs who have lower levels of intervention integrity or who have significant drift are provided detailed feedback and supervision.

3c) Participant recruitment and randomization: The 20 selected clinics are randomly assigned into 5 clusters (4 clusters of 4 clinics from the same city and 1 cluster of 4 clinics from two cities). In each cluster, CBO members and health care staff distribute flyers and CBO members working in each MMT clinic approach patients when patients come daily for their MMT dosages to invite them to participate in self-screening with tablet-based ASSIST as well as urine drug test and Quick HIV tests. Once agreed, CBO assist with self-screening processes. Individuals who participate in self-screening give verbal agreement to participate and receive compensation for their time. Those with low-risk scores and urine negative with meth metabolites are offered a Brief Intervention by trained CBO members. Those with reactive Quick HIV tests are referred to HIV care facilities if these participants have not done so.

Recruiting participants for adaptive interventions:

CBO members invite those who are at moderate-risk and high-risk scores for meth or have urine positive with meth metabolites to participate in the study. Those who express interest and provide contact information are referred to research assistants (RA) who then makes appointment to screen for eligibility. At each clinic, RA conduct a brief survey and collect urine sample to confirm recent meth use. The study over-recruits women as the majority of MMT patients in Vietnam are men. The study aims to recruit 200 HIV+ and 400 HIV-. Those who sign informed consent are enrolled in baseline assessment and electronically fingerprinted to create unique ID. Participants receive compensation for their participation in baseline assessment. Eligible participants at each clinic are first stratified by HIV status, and then randomized to low vs. high intensity frontline interventions.

4) Cost-effectiveness analysis of interventions (Aim 2) 4a) The cost-effectiveness analysis has two goals: 1) to determine whether any additional improvement in outcomes associated with interventions of different intensity and expense is worth the additional cost; and 2) to provide guidance to the Vietnam Ministry of Health on the cost of scaling-up and implementing the interventions. This analysis measures the increment in cost between contrasted interventions divided by the increment in outcomes. Effectiveness of each intervention for HIV+ and HIV- groups is measured by the estimated outcome probabilities for each outcome of interest, as in Aim 1.

4b) Costs are assessed from the point of view of the public health agency. The second analysis will include social costs. Implementation costs are calculated based on costs for each arm incurred by health care providers, including costs of implementing the intervention, mental health and drug treatment services used. An activity-based costing approach is used to estimate the cost of fielding the interventions in 20 MMT clinics. A template is used to collect data on salaries for personnel and consultants, physical resources, clinical supplies and miscellaneous charges that are required to deliver each intervention type. Data is collected from participants on medical visits and involvement with the criminal justice system. These differences are costed out using local pricing data. Per capita costs for each intervention are calculated by dividing the total cost for each site/arm by the number of participants in each arm at that site.

5) Ethnographic evaluation to identify the structural, provider, and patient-level factors that influence adoption and scale-up of interventions in MMT clinics. (Aim 3).

5a) Ethnographic interviews: Two ethnographic researchers conduct pre-post intervention in-depth interviews with 12 individuals in each cluster of clinics. Participants include MMT manager, MMT clinical staff, CBO members and patients who participate in interventions. In each cluster, at least 6 patients are selected. In-depth ethnographic interviews with these individuals take place immediately before enrollment and immediately after maintenance or enhanced treatments end.

With CBO and MMT staff, pre-intervention interviews explore experiences with current work; experiences with meth users, expectations of whether and how the interventions would work. Post-intervention interviews explore actual experiences with delivering interventions as well as perceived barriers and facilitators for adoption and scale-up.

With participants: first interviews explore family of origin, childhood and coming of age; histories of sexual and affective relations; histories of drug use and patterns of meth use; current social support; broader life goals; motivations to participate in the study, and expectations of how the interventions would work. Second interviews explore actual experiences and outcomes as well as motivations to stay in the interventions.

The Consolidated Framework for Implementation Research is used in all interviews to probe participant perceptions of the characteristics of the STAR-OM interventions, of outer settings, inner settings, provider characteristics and the implementation process.

5b) Ethnographic Observation: Two kinds of observations take place. The first, carried out with in-depth interviews of participants who consent to participate in this additional form of data collection, involves having two ethnographers spend time with them to observe activities such as individual meetings, group activities and other daily activities in the clinical and/or community settings. The second element of observation involve Master Counselors to observe randomly selected sessions of interventions in CM and CBT period and keep a logbook of SMS messages that are sent out to each participant in the study. A checklist is used to assess the fidelity of interventions contents and delivery. Master Counselors also assess other contextual information that is useful to determine whether interventions are effectively delivered. All observation periods are recorded with detailed field notes.

ELIGIBILITY:
Inclusion Criteria:

* ASSIST scores from 10+ for methamphetamine use OR Confirmed methamphetamine use with urine analysis;
* Willing to provide at least three pieces of contact information;
* Having a cell phone to receive texts.

Exclusion Criteria:

* Psychosis or other interfering problems;
* Cannot understand study procedures as judged by research assistants.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Le Minh Giang, PhD, Principal Investigator — Hanoi Medical University; Steve Shoptaw, PhD, Principal Investigator — University of California, Los Angeles, Department of Family Medicine
Locations (4):
- Vietnam (4):
  - Hai Ba Trung methadone clinic, Hanoi, Hanoi
  - Long Bien methadone clinic, Hanoi, Hanoi
  - Nam Tu Liem Methadone clinic, Hanoi, Hanoi
  - District 4 Methadone clinic, Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Nguyen TT, Nguyen LT, Pham MD, Vu HH, Mulvey KP. Methadone maintenance therapy in Vietnam: an overview and scaling-up plan. Adv Prev Med. 2012;2012:732484. doi: 10.1155/2012/732484. Epub 2012 Nov 25. PMID 23227351
- [Background] Des Jarlais DC, Thi Huong D, Thi Hai Oanh K, Khue Pham M, Thi Giang H, Thi Tuyet Thanh N, Arasteh K, Feelemyer J, Hammett T, Peries M, Michel L, Vu Hai V, Roustide MJ, Moles JP, Laureillard D, Nagot N; DRIVE Study Team. Prospects for ending the HIV epidemic among persons who inject drugs in Haiphong, Vietnam. Int J Drug Policy. 2016 Jun;32:50-6. doi: 10.1016/j.drugpo.2016.02.021. Epub 2016 Feb 27. PMID 27006257
- [Background] Giang L, Thuy D, Trang N, Okafor CN, Li M, Shoptaw S. Severity of methamphetamine use among methadone patients in Vietnam: Prevalence and correlates (Poster presentation at CPDD 81st Annual Scientific Meeting). San Antonio, Texas; 2019
- [Background] Vietnam Ministry of Health. Báo cáo Đánh giá và tổng kết 10 năm triển khai chương trình điều trị nghiện các chất dạng thuốc phiện bằng thuốc Methadone (Assessment and Review of 10 Years of Methadone Maintenance Therapy in Vietnam: Report to the Prime Minister) (DRAFT). Vietnam Ministry of Health; n.d.
- [Background] Feelemyer J, Duong Thi H, Khue Pham M, Hoang Thi G, Thi Tuyet Thanh N, Thi Hai Oanh K, Arasteh K, Moles JP, Vu Hai V, Vallo R, Quillet C, Rapoud D, Michel L, Hammett T, Laureillard D, Nagot N, Des Jarlais D; DRIVE Study Team. Increased Methamphetamine Use among Persons Who Inject Drugs in Hai Phong, Vietnam, and the Association with Injection and Sexual Risk Behaviors. J Psychoactive Drugs. 2018 Nov-Dec;50(5):382-389. doi: 10.1080/02791072.2018.1508790. Epub 2018 Sep 5. PMID 30183558
- [Background] Korthuis PT, Bart G, Kunkel LE, Diep NB, Brinkerhoff C, Giang LM. Buprenorphine versus Methadone impact on the HIV care continuum in Vietnam: BRAVCO study 6-month outcomes (Poster presentation at 79th CPDD Annual Scientific Meeting). San Diego, CA; 2018.
- [Background] Ellis MS, Kasper ZA, Cicero TJ. Twin epidemics: The surging rise of methamphetamine use in chronic opioid users. Drug Alcohol Depend. 2018 Dec 1;193:14-20. doi: 10.1016/j.drugalcdep.2018.08.029. Epub 2018 Oct 10. PMID 30326396
- [Background] Shariatirad S, Maarefvand M, Ekhtiari H. Methamphetamine use and methadone maintenance treatment: an emerging problem in the drug addiction treatment network in Iran. Int J Drug Policy. 2013 Nov;24(6):e115-6. doi: 10.1016/j.drugpo.2013.05.003. Epub 2013 Jun 15. No abstract available. PMID 23773684
- [Background] Wang R, Ding Y, Bai H, Duan S, Ye R, Yang Y, Wang J, Tang R, Gao M, He N. Illicit Heroin and Methamphetamine Use among Methadone Maintenance Treatment Patients in Dehong Prefecture of Yunnan Province, China. PLoS One. 2015 Jul 21;10(7):e0133431. doi: 10.1371/journal.pone.0133431. eCollection 2015. PMID 26196394
- [Background] Al-Tayyib A, Koester S, Langegger S, Raville L. Heroin and Methamphetamine Injection: An Emerging Drug Use Pattern. Subst Use Misuse. 2017 Jul 3;52(8):1051-1058. doi: 10.1080/10826084.2016.1271432. Epub 2017 Mar 21. PMID 28323507
- [Background] Parsons JT, John SA, Millar BM, Starks TJ. Testing the Efficacy of Combined Motivational Interviewing and Cognitive Behavioral Skills Training to Reduce Methamphetamine Use and Improve HIV Medication Adherence Among HIV-Positive Gay and Bisexual Men. AIDS Behav. 2018 Aug;22(8):2674-2686. doi: 10.1007/s10461-018-2086-5. PMID 29536284
- [Background] Huang YS, Tang TC, Lin CH, Yen CF. Effects of motivational enhancement therapy on readiness to change MDMA and methamphetamine use behaviors in Taiwanese adolescents. Subst Use Misuse. 2011;46(4):411-6. doi: 10.3109/10826084.2010.501664. Epub 2010 Aug 24. PMID 20735217
- [Background] Galloway GP, Polcin D, Kielstein A, Brown M, Mendelson J. A nine session manual of motivational enhancement therapy for methamphetamine dependence: adherence and efficacy. J Psychoactive Drugs. 2007 Nov;Suppl 4:393-400. doi: 10.1080/02791072.2007.10399900. PMID 18286727
- [Background] Lee NK, Rawson RA. A systematic review of cognitive and behavioural therapies for methamphetamine dependence. Drug Alcohol Rev. 2008 May;27(3):309-17. doi: 10.1080/09595230801919494. PMID 18368613
- [Background] Rajasingham R, Mimiaga MJ, White JM, Pinkston MM, Baden RP, Mitty JA. A systematic review of behavioral and treatment outcome studies among HIV-infected men who have sex with men who abuse crystal methamphetamine. AIDS Patient Care STDS. 2012 Jan;26(1):36-52. doi: 10.1089/apc.2011.0153. Epub 2011 Nov 9. PMID 22070609
- [Background] Reback CJ, Peck JA, Dierst-Davies R, Nuno M, Kamien JB, Amass L. Contingency management among homeless, out-of-treatment men who have sex with men. J Subst Abuse Treat. 2010 Oct;39(3):255-63. doi: 10.1016/j.jsat.2010.06.007. Epub 2010 Jul 29. PMID 20667681
- [Background] Menza TW, Jameson DR, Hughes JP, Colfax GN, Shoptaw S, Golden MR. Contingency management to reduce methamphetamine use and sexual risk among men who have sex with men: a randomized controlled trial. BMC Public Health. 2010 Dec 20;10:774. doi: 10.1186/1471-2458-10-774. PMID 21172026
- [Background] Rawson RA, McCann MJ, Flammino F, Shoptaw S, Miotto K, Reiber C, Ling W. A comparison of contingency management and cognitive-behavioral approaches for stimulant-dependent individuals. Addiction. 2006 Feb;101(2):267-74. doi: 10.1111/j.1360-0443.2006.01312.x. PMID 16445555
- [Background] Rawson RA, Marinelli-Casey P, Anglin MD, Dickow A, Frazier Y, Gallagher C, Galloway GP, Herrell J, Huber A, McCann MJ, Obert J, Pennell S, Reiber C, Vandersloot D, Zweben J; Methamphetamine Treatment Project Corporate Authors. A multi-site comparison of psychosocial approaches for the treatment of methamphetamine dependence. Addiction. 2004 Jun;99(6):708-17. doi: 10.1111/j.1360-0443.2004.00707.x. PMID 15139869
- [Background] Carrico AW, Flentje A, Gruber VA, Woods WJ, Discepola MV, Dilworth SE, Neilands TB, Jain J, Siever MD. Community-based harm reduction substance abuse treatment with methamphetamine-using men who have sex with men. J Urban Health. 2014 Jun;91(3):555-67. doi: 10.1007/s11524-014-9870-y. PMID 24744105
- [Background] Magidson JF, Gouse H, Burnhams W, Wu CY, Myers B, Joska JA, Carrico AW. Beyond methamphetamine: Documenting the implementation of the Matrix model of substance use treatment for opioid users in a South African setting. Addict Behav. 2017 Mar;66:132-137. doi: 10.1016/j.addbeh.2016.11.014. Epub 2016 Nov 17. PMID 27940387
- [Background] Reback CJ, Fletcher JB, Leibowitz AA. Cost effectiveness of text messages to reduce methamphetamine use and HIV sexual risk behaviors among men who have sex with men. J Subst Abuse Treat. 2019 May;100:59-63. doi: 10.1016/j.jsat.2019.02.006. Epub 2019 Feb 27. PMID 30898329
- [Background] Reback CJ, Fletcher JB, Swendeman DA, Metzner M. Theory-Based Text-Messaging to Reduce Methamphetamine Use and HIV Sexual Risk Behaviors Among Men Who Have Sex with Men: Automated Unidirectional Delivery Outperforms Bidirectional Peer Interactive Delivery. AIDS Behav. 2019 Jan;23(1):37-47. doi: 10.1007/s10461-018-2225-z. PMID 30006792
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Degenhardt L, Mathers B, Guarinieri M, Panda S, Phillips B, Strathdee SA, Tyndall M, Wiessing L, Wodak A, Howard J; Reference Group to the United Nations on HIV and injecting drug use. Meth/amphetamine use and associated HIV: Implications for global policy and public health. Int J Drug Policy. 2010 Sep;21(5):347-58. doi: 10.1016/j.drugpo.2009.11.007. Epub 2010 Feb 1. PMID 20117923
- [Background] UNODC. World Drug Report 2018. Vienna, Austria: United Nations Ofice on Drugs and Crime; 2018
- [Background] Colfax G, Santos GM, Chu P, Vittinghoff E, Pluddemann A, Kumar S, Hart C. Amphetamine-group substances and HIV. Lancet. 2010 Aug 7;376(9739):458-74. doi: 10.1016/S0140-6736(10)60753-2. PMID 20650520
- [Background] Gonzales R, Mooney L, Rawson RA. The methamphetamine problem in the United States. Annu Rev Public Health. 2010;31:385-98. doi: 10.1146/annurev.publhealth.012809.103600. PMID 20070191
- [Background] Strathdee SA, Stockman JK. Epidemiology of HIV among injecting and non-injecting drug users: current trends and implications for interventions. Curr HIV/AIDS Rep. 2010 May;7(2):99-106. doi: 10.1007/s11904-010-0043-7. PMID 20425564
- [Background] Conners EE, Gaines TL, Strathdee SA, Magis-Rodriguez C, Brouwer KC. Structural factors associated with methamphetamine smoking among female sex workers in Tijuana, Mexico. Drug Alcohol Rev. 2018 Apr;37 Suppl 1(Suppl 1):S294-S302. doi: 10.1111/dar.12633. Epub 2017 Dec 7. PMID 29218799
- [Background] García-Aurrecoechea VR, Gutiérrez-López AD, Rodríguez-Kuri SE, Velázquez-Altamirano M, Fernández-Cáceres C. Increasing methamphetamine use trends alert among patients in Mexico. J Subst Use. 2018 Feb 5;0(0):1-6.
- [Background] Liu D, Jiang Z, Xiu C, Li Z, Song Q, Wang Z. Sexually transmitted infection prevalence and related risk factors among heterosexual male methamphetamine users in China. Int J STD AIDS. 2017 Oct;28(12):1208-1214. doi: 10.1177/0956462417693165. Epub 2017 Feb 8. PMID 28178893
- [Background] Liao M, Kang D, Tao X, Li J, Qian Y, Wang G, Jiang B, Bi Z, Jia Y. Dual epidemics of syphilis and methamphetamine use among drug users in Shandong Province of China. AIDS Care. 2013;25(10):1236-44. doi: 10.1080/09540121.2013.764384. Epub 2013 Feb 11. PMID 23394142
- [Background] Celentano DD, Sirirojn B, Sutcliffe CG, Quan VM, Thomson N, Keawvichit R, Wongworapat K, Latkin C, Taechareonkul S, Sherman SG, Aramrattana A. Sexually transmitted infections and sexual and substance use correlates among young adults in Chiang Mai, Thailand. Sex Transm Dis. 2008 Apr;35(4):400-5. doi: 10.1097/OLQ.0b013e31815fd412. PMID 18362863
- [Background] Beyrer C, Razak MH, Jittiwutikarn J, Suriyanon V, Vongchak T, Srirak N, Kawichai S, Tovanabutra S, Rungruengthanakit K, Sawanpanyalert P, Sripaipan T, Celentano DD. Methamphetamine users in northern Thailand: changing demographics and risks for HIV and STD among treatment-seeking substance abusers. Int J STD AIDS. 2004 Oct;15(10):697-704. doi: 10.1177/095646240401501012. PMID 15479508
- [Background] Prybylski D, Manopaiboon C, Visavakum P, Yongvanitjit K, Aramrattana A, Manomaipiboon P, Tanpradech S, Suksripanich O, Pattanasin S, Wolfe M, Whitehead SJ. Diverse HIV epidemics among people who inject drugs in Thailand: evidence from respondent-driven sampling surveys in Bangkok and Chiang Mai. Drug Alcohol Depend. 2015 Mar 1;148:126-35. doi: 10.1016/j.drugalcdep.2014.12.034. Epub 2015 Jan 12. PMID 25640153
- [Background] Morris K, Parry C. South African methamphetamine boom could fuel further HIV. Lancet Infect Dis. 2006 Aug;6(8):471. doi: 10.1016/s1473-3099(06)70539-4. No abstract available. PMID 16888875
- [Background] Gouse H, Joska JA, Lion RR, Watt MH, Burnhams W, Carrico AW, Meade CS. HIV testing and sero-prevalence among methamphetamine users seeking substance abuse treatment in Cape Town. Drug Alcohol Rev. 2016 Sep;35(5):580-3. doi: 10.1111/dar.12371. Epub 2015 Dec 14. PMID 26661781
- [Background] Shoptaw S, Reback CJ. Methamphetamine use and infectious disease-related behaviors in men who have sex with men: implications for interventions. Addiction. 2007 Apr;102 Suppl 1:130-5. doi: 10.1111/j.1360-0443.2006.01775.x. PMID 17493062
- [Background] Garofalo R, Mustanski BS, McKirnan DJ, Herrick A, Donenberg GR. Methamphetamine and young men who have sex with men: understanding patterns and correlates of use and the association with HIV-related sexual risk. Arch Pediatr Adolesc Med. 2007 Jun;161(6):591-6. doi: 10.1001/archpedi.161.6.591. PMID 17548765
- [Background] Wu H, Xiu C, Fu X, Li M, Wang Z, Li X, Wu J, Vermund SH, Hu Y. Syphilis associated with recreational drug use, depression and high-risk sexual behaviour in men who have sex with men: a case-control study in China. Sex Transm Infect. 2019 Jun;95(4):267-272. doi: 10.1136/sextrans-2018-053878. Epub 2019 Mar 6. PMID 30842346
- [Background] Nerlander LMC, Hoots BE, Bradley H, Broz D, Thorson A, Paz-Bailey G; NHBS Group. HIV infection among MSM who inject methamphetamine in 8 US cities. Drug Alcohol Depend. 2018 Sep 1;190:216-223. doi: 10.1016/j.drugalcdep.2018.06.017. Epub 2018 Jul 20. PMID 30055426
- [Background] Vu NT, Holt M, Phan HT, La LT, Tran GM, Doan TT, Nguyen TN, de Wit J. The Relationship Between Methamphetamine Use, Sexual Sensation Seeking and Condomless Anal Intercourse Among Men Who Have Sex With Men in Vietnam: Results of a Community-Based, Cross-Sectional Study. AIDS Behav. 2017 Apr;21(4):1105-1116. doi: 10.1007/s10461-016-1467-x. PMID 27351193
- [Background] Jin H, Ogunbajo A, Mimiaga MJ, Duncan DT, Boyer E, Chai P, Dilworth SE, Carrico AW. Over the influence: The HIV care continuum among methamphetamine-using men who have sex with men. Drug Alcohol Depend. 2018 Nov 1;192:125-128. doi: 10.1016/j.drugalcdep.2018.07.038. Epub 2018 Sep 13. PMID 30248558
- [Background] Moore DJ, Blackstone K, Woods SP, Ellis RJ, Atkinson JH, Heaton RK, Grant I; Hnrc Group And The Tmarc Group. Methamphetamine use and neuropsychiatric factors are associated with antiretroviral non-adherence. AIDS Care. 2012;24(12):1504-13. doi: 10.1080/09540121.2012.672718. Epub 2012 Apr 24. PMID 22530794
- [Background] Feldman MB, Kepler KL, Irvine MK, Thomas JA. Associations between drug use patterns and viral load suppression among HIV-positive individuals who use support services in New York City. Drug Alcohol Depend. 2019 Apr 1;197:15-21. doi: 10.1016/j.drugalcdep.2018.12.015. Epub 2019 Jan 15. PMID 30743195
- [Background] Aralis HJ, Shoptaw S, Brookmeyer R, Ragsdale A, Bolan R, Gorbach PM. Psychiatric Illness, Substance Use, and Viral Suppression Among HIV-Positive Men of Color Who Have Sex with Men in Los Angeles. AIDS Behav. 2018 Oct;22(10):3117-3129. doi: 10.1007/s10461-018-2055-z. PMID 29478146
- [Background] Hojilla JC, Vlahov D, Glidden DV, Amico KR, Mehrotra M, Hance R, Grant RM, Carrico AW. Skating on thin ice: stimulant use and sub-optimal adherence to HIV pre-exposure prophylaxis. J Int AIDS Soc. 2018 Mar;21(3):e25103. doi: 10.1002/jia2.25103. PMID 29577616
- [Background] Grov C, Rendina HJ, John SA, Parsons JT. Determining the Roles that Club Drugs, Marijuana, and Heavy Drinking Play in PrEP Medication Adherence Among Gay and Bisexual Men: Implications for Treatment and Research. AIDS Behav. 2019 May;23(5):1277-1286. doi: 10.1007/s10461-018-2309-9. PMID 30306433
- [Background] Carrico AW, Flentje A, Kober K, Lee S, Hunt P, Riley ED, Shoptaw S, Flowers E, Dilworth SE, Pahwa S, Aouizerat BE. Recent stimulant use and leukocyte gene expression in methamphetamine users with treated HIV infection. Brain Behav Immun. 2018 Jul;71:108-115. doi: 10.1016/j.bbi.2018.04.004. Epub 2018 Apr 18. PMID 29679637
- [Background] Carrico AW, Cherenack EM, Roach ME, Riley ED, Oni O, Dilworth SE, Shoptaw S, Hunt P, Roy S, Pallikkuth S, Pahwa S. Substance-associated elevations in monocyte activation among methamphetamine users with treated HIV infection. AIDS. 2018 Mar 27;32(6):767-771. doi: 10.1097/QAD.0000000000001751. PMID 29369159
- [Background] Daniulaityte R, Juhascik MP, Strayer KE, Sizemore IE, Zatreh M, Nahhas RW, Harshbarger KE, Antonides HM, Martins SS, Carlson RG. Trends in fentanyl and fentanyl analogue-related overdose deaths - Montgomery County, Ohio, 2015-2017. Drug Alcohol Depend. 2019 May 1;198:116-120. doi: 10.1016/j.drugalcdep.2019.01.045. Epub 2019 Mar 18. PMID 30909018
- [Background] Robles F. Meth, the Forgotten Killer, Is Back. And It's Everywhere. N Y Times [Internet]. 2018 Feb 15 [cited 2019 Apr 28]; Available from: https://www.nytimes.com/2018/02/13/us/meth-crystal-drug.html
- [Background] Magill M, Ray LA. Cognitive-behavioral treatment with adult alcohol and illicit drug users: a meta-analysis of randomized controlled trials. J Stud Alcohol Drugs. 2009 Jul;70(4):516-27. doi: 10.15288/jsad.2009.70.516. PMID 19515291
- [Background] Benishek LA, Dugosh KL, Kirby KC, Matejkowski J, Clements NT, Seymour BL, Festinger DS. Prize-based contingency management for the treatment of substance abusers: a meta-analysis. Addiction. 2014 Sep;109(9):1426-36. doi: 10.1111/add.12589. Epub 2014 May 23. PMID 24750232
- [Background] Dutra L, Stathopoulou G, Basden SL, Leyro TM, Powers MB, Otto MW. A meta-analytic review of psychosocial interventions for substance use disorders. Am J Psychiatry. 2008 Feb;165(2):179-87. doi: 10.1176/appi.ajp.2007.06111851. Epub 2008 Jan 15. PMID 18198270
- [Background] Prendergast M, Podus D, Finney J, Greenwell L, Roll J. Contingency management for treatment of substance use disorders: a meta-analysis. Addiction. 2006 Nov;101(11):1546-60. doi: 10.1111/j.1360-0443.2006.01581.x. PMID 17034434
- [Background] Carroll KM. Lost in translation? Moving contingency management and cognitive behavioral therapy into clinical practice. Ann N Y Acad Sci. 2014 Oct;1327(1):94-111. doi: 10.1111/nyas.12501. Epub 2014 Sep 9. PMID 25204847
- [Background] Nguyen Huu C, Kieu Cong T. Application of Matrix model in support of trreatment and recovery for ATS dependents (Nghiên cứu sử dụng liệu pháp tâm lý Matrix trong hỗ trợ điều trị nghiện và phục hồi chức năng cho người nghiện ma túy tổng hợp dạng amphetamine). Conference Presentation presented at: Treatment Approaches for ATS Dependence; 2016 Dec 20; Hanoi, Vietnam
- [Background] Giang L, Thuy D, Trang N, Okafor CN, Li M, Shoptaw S. Feasibility And Outcomes Of Evidence-Based Interventions To Reduce Methamphetamine Use Among Patients On Methadone Maintenance Therapy In Hanoi, Vietnam (Poster presentation at 2019 NIDA International Forum). San Antonio, Texas; 2019.
- [Background] Young MM, Stevens A, Porath-Waller A, Pirie T, Garritty C, Skidmore B, Turner L, Arratoon C, Haley N, Leslie K, Reardon R, Sproule B, Grimshaw J, Moher D. Effectiveness of brief interventions as part of the screening, brief intervention and referral to treatment (SBIRT) model for reducing the non-medical use of psychoactive substances: a systematic review protocol. Syst Rev. 2012 May 7;1:22. doi: 10.1186/2046-4053-1-22. PMID 22587894
- [Background] Reavis-Scruggs R, Wilder AD. An alternative method for polishing amalgam restorations. Dent Hyg (Chic). 1985 Oct;59(10):458-60. No abstract available. PMID 3865817
- [Background] Gelberg L, Andersen RM, Afifi AA, Leake BD, Arangua L, Vahidi M, Singleton K, Yacenda-Murphy J, Shoptaw S, Fleming MF, Baumeister SE. Project QUIT (Quit Using Drugs Intervention Trial): a randomized controlled trial of a primary care-based multi-component brief intervention to reduce risky drug use. Addiction. 2015 Nov;110(11):1777-90. doi: 10.1111/add.12993. PMID 26471159
- [Background] Baumeister SE, Gelberg L, Leake BD, Yacenda-Murphy J, Vahidi M, Andersen RM. Effect of a primary care based brief intervention trial among risky drug users on health-related quality of life. Drug Alcohol Depend. 2014 Sep 1;142:254-61. doi: 10.1016/j.drugalcdep.2014.06.034. Epub 2014 Jul 4. PMID 25042213
- [Background] Reback CJ, Fletcher JB, Shoptaw S, Mansergh G. Exposure to Theory-Driven Text Messages is Associated with HIV Risk Reduction Among Methamphetamine-Using Men Who have Sex with Men. AIDS Behav. 2015 Jun;19 Suppl 2:130-41. doi: 10.1007/s10461-014-0985-7. PMID 25563501
- [Background] Gomicronmez W, Olem D, Andrews R, Discepola MV, Ambrose P, Dilworth SE, Carrico AW. Optimizing Contingency Management with Methamphetamine-Using Men who Have Sex with Men. Cogn Behav Pract. 2018 May;25(2):286-295. doi: 10.1016/j.cbpra.2017.08.003. Epub 2017 Sep 11. PMID 32461714
- [Background] Charoenlarp P, Radomyos P. Treatment of Raillietina siriraji with atabrine. Southeast Asian J Trop Med Public Health. 1973 Jun;4(2):288. No abstract available. PMID 4795974
- [Background] Amato L, Minozzi S, Davoli M, Vecchi S. Psychosocial combined with agonist maintenance treatments versus agonist maintenance treatments alone for treatment of opioid dependence. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD004147. doi: 10.1002/14651858.CD004147.pub4. PMID 21975742
- [Background] UNODC. The Challenge of Synthetic Drugs in East and South-East Asia and Oceania: Trends and Patterns of Amphetamine-type Stimulants and New Psychoactive Substances. Vienna, Austria: United Nations Office on Drugs and Crime; 2015 May.
- [Background] Bao YP, Liu ZM, Li JH, Zhang RM, Hao W, Zhao M, Shi J, McGoogan JM, Lu L. Club drug use and associated high-risk sexual behaviour in six provinces in China. Addiction. 2015 Jan;110 Suppl 1:11-9. doi: 10.1111/add.12770. PMID 25533860
- [Background] Carrico AW, Nil E, Sophal C, Stein E, Sokunny M, Yuthea N, Evans JL, Ngak S, Maher L, Page K. Behavioral interventions for Cambodian female entertainment and sex workers who use amphetamine-type stimulants. J Behav Med. 2016 Jun;39(3):502-10. doi: 10.1007/s10865-016-9713-2. Epub 2016 Jan 18. PMID 26782667
- [Background] Zhang C, Liu Y, Sun X, Wang J, Lu HY, He X, Zhang H, Ruan YH, Shao Y, Vermund SH, Qian HZ. Substance use and HIV-risk behaviors among HIV-positive men who have sex with men in China: repeated measures in a cohort study design. AIDS Care. 2017 May;29(5):644-653. doi: 10.1080/09540121.2016.1255709. Epub 2016 Nov 10. PMID 27832699
- [Background] Liu D, Gu J, Xu H, Hao C, Jiao M, Zhang X, Zhao Y, Andrew B, Hao Y. Club drugs and alcohol abuse predicted dropout and poor adherence among methadone maintenance treatment patients in Guangzhou, China. AIDS Care. 2017 Apr;29(4):458-463. doi: 10.1080/09540121.2016.1259452. Epub 2016 Nov 30. PMID 27903083
- [Background] Alam-mehrjerdi Z, Mokri A, Dolan K. Methamphetamine use and treatment in Iran: A systematic review from the most populated Persian Gulf country. Asian J Psychiatr. 2015 Aug;16:17-25. doi: 10.1016/j.ajp.2015.05.036. Epub 2015 May 28. PMID 26123235
- [Background] Watt MH, Meade CS, Kimani S, MacFarlane JC, Choi KW, Skinner D, Pieterse D, Kalichman SC, Sikkema KJ. The impact of methamphetamine ("tik") on a peri-urban community in Cape Town, South Africa. Int J Drug Policy. 2014 Mar;25(2):219-25. doi: 10.1016/j.drugpo.2013.10.007. Epub 2013 Oct 26. PMID 24246503
- [Background] Petersen I, Evans-Lacko S, Semrau M, Barry MM, Chisholm D, Gronholm P, Egbe CO, Thornicroft G. Promotion, prevention and protection: interventions at the population- and community-levels for mental, neurological and substance use disorders in low- and middle-income countries. Int J Ment Health Syst. 2016 Apr 11;10:30. doi: 10.1186/s13033-016-0060-z. eCollection 2016. PMID 27069506
- [Background] Baingana F, al'Absi M, Becker AE, Pringle B. Global research challenges and opportunities for mental health and substance-use disorders. Nature. 2015 Nov 19;527(7578):S172-7. doi: 10.1038/nature16032. PMID 26580324
- [Background] Assanangkornchai S, Balthip Q, Edwards JG; assistance of the ASSIST-SBI Development Co-investigators. Implementing the Alcohol, Smoking, Substance Involvement Screening Test and linked brief intervention service in primary care in Thailand. J Public Health (Oxf). 2014 Sep;36(3):443-9. doi: 10.1093/pubmed/fdu011. Epub 2014 Feb 25. PMID 24573365
- [Background] Wechsberg WM, Luseno WK, Karg RS, Young S, Rodman N, Myers B, Parry CD. Alcohol, cannabis, and methamphetamine use and other risk behaviours among Black and Coloured South African women: a small randomized trial in the Western Cape. Int J Drug Policy. 2008 Apr;19(2):130-9. doi: 10.1016/j.drugpo.2007.11.018. Epub 2008 Jan 18. PMID 18207723
- [Background] Sorsdahl K, Myers B, Ward C, Matzopoulos R, Mtukushe B, Nicol A, Stein DJ. Screening and brief interventions for substance use in emergency departments in the Western Cape province of South Africa: views of health care professionals. Int J Inj Contr Saf Promot. 2014;21(3):236-43. doi: 10.1080/17457300.2013.811267. Epub 2013 Jul 9. PMID 23837749
- [Background] Hser YI, Li J, Jiang H, Zhang R, Du J, Zhang C, Zhang B, Evans E, Wu F, Chang YJ, Peng C, Huang D, Stitzer ML, Roll J, Zhao M. Effects of a randomized contingency management intervention on opiate abstinence and retention in methadone maintenance treatment in China. Addiction. 2011 Oct;106(10):1801-9. doi: 10.1111/j.1360-0443.2011.03490.x. Epub 2011 Jul 27. PMID 21793958
- [Background] Chen W, Hong Y, Zou X, McLaughlin MM, Xia Y, Ling L. Effectiveness of prize-based contingency management in a methadone maintenance program in China. Drug Alcohol Depend. 2013 Nov 1;133(1):270-4. doi: 10.1016/j.drugalcdep.2013.05.028. Epub 2013 Jul 4. PMID 23831409
- [Background] Cohen A, Riley D, McGregor C. The Emergence of Methamphetamine in Thailand: Interventions and Treatment. In: Pates R, Riley D, editors. Interv Amphetamine Misuse. Oxford, UK: John Wiley & Sons; 2009. p. 159-172.
- [Background] Rawson RA, Huber A, McCann M, Shoptaw S, Farabee D, Reiber C, Ling W. A comparison of contingency management and cognitive-behavioral approaches during methadone maintenance treatment for cocaine dependence. Arch Gen Psychiatry. 2002 Sep;59(9):817-24. doi: 10.1001/archpsyc.59.9.817. PMID 12215081
- [Background] Roux P, Lions C, Vilotitch A, Michel L, Mora M, Maradan G, Marcellin F, Spire B, Morel A, Carrieri PM; ANRS Methaville study group. Correlates of cocaine use during methadone treatment: implications for screening and clinical management (ANRS Methaville study). Harm Reduct J. 2016 Apr 5;13:12. doi: 10.1186/s12954-016-0100-7. PMID 27048152
- [Background] Giang LM, Ngoc LB, Hoang VH, Mulvey K, Rawson RA. Substance use disorders and HIV in Vietnam since Doi Moi (Renovation): an overview. J Food Drug Anal. 2013 Dec;21(4):S42-S45. doi: 10.1016/j.jfda.2013.09.032. PMID 25278736
- [Background] Ho HT, Le GM, Dinh TT. Female sex workers who use amphetamine-type stimulants (ATS) in three cities of Vietnam: use and sexual risks related to HIV/AIDS. Glob Public Health. 2013;8(5):552-69. doi: 10.1080/17441692.2013.790459. Epub 2013 May 16. PMID 23679831
- [Background] Yu G, Clatts MC, Goldsamt LA, Giang le M. Substance use among male sex workers in Vietnam: prevalence, onset, and interactions with sexual risk. Int J Drug Policy. 2015 May;26(5):516-21. doi: 10.1016/j.drugpo.2014.10.011. Epub 2014 Nov 8. PMID 25488636
- [Background] Vuong T, Shanahan M, Nguyen N, Le G, Ali R, Pham K, Vuong TTA, Dinh T, Ritter A. Cost-effectiveness of center-based compulsory rehabilitation compared to community-based voluntary methadone maintenance treatment in Hai Phong City, Vietnam. Drug Alcohol Depend. 2016 Nov 1;168:147-155. doi: 10.1016/j.drugalcdep.2016.09.008. Epub 2016 Sep 13. PMID 27664552
- [Background] Nguyen Bich D, Korthuis PT, Nguyen Thu T, Van Dinh H, Le Minh G. HIV Patients' Preference for Integrated Models of Addiction and HIV Treatment in Vietnam. J Subst Abuse Treat. 2016 Oct;69:57-63. doi: 10.1016/j.jsat.2016.07.003. Epub 2016 Jul 19. PMID 27568511
- [Background] Clatts MC, Goldsamt LA, Giang LM, Quoc Bao L, Yu G, Colby D. Sexually transmissible infection and HIV prevention and treatment for young male sex workers in Vietnam: findings from the SHEATH intervention. Sex Health. 2016 Nov;13(6):575-581. doi: 10.1071/SH16051. PMID 27607764
- [Background] Clatts MC, Goldsamt LA, Giang le M, Yu G. Sexual practices, partner concurrency and high rates of sexually transmissible infections among male sex workers in three cities in Vietnam. Sex Health. 2015 Mar;12(1):39-47. doi: 10.1071/SH14101. PMID 25622225
- [Background] Nguyen TT, Luong AN, Nham TTT, Chauvin C, Feelemyer J, Nagot N, Jarlais DD, Le MG, Jauffret-Roustide M. Struggling to achieve a 'normal life': A qualitative study of Vietnamese methadone patients. Int J Drug Policy. 2019 Jun;68:18-26. doi: 10.1016/j.drugpo.2019.03.026. Epub 2019 Apr 9. PMID 30978641
- [Background] Carrico AW, Jain J, Discepola MV, Olem D, Andrews R, Woods WJ, Neilands TB, Shoptaw S, Gomez W, Dilworth SE, Moskowitz JT. A community-engaged randomized controlled trial of an integrative intervention with HIV-positive, methamphetamine-using men who have sex with men. BMC Public Health. 2016 Jul 30;16:673. doi: 10.1186/s12889-016-3325-1. PMID 27476110
- [Background] Worley MJ, Swanson A-N, Heinzerling KG, Roche DJ, Shoptaw S. Ibudilast attenuates subjective effects of methamphetamine in a placebo-controlled inpatient study. Drug Alcohol Depend. 2016 May 1;162:245-50. doi: 10.1016/j.drugalcdep.2016.02.036. Epub 2016 Mar 3. PMID 26993372
- [Background] Shoptaw S, Watson DW, Reiber C, Rawson RA, Montgomery MA, Majewska MD, Ling W. Randomized controlled pilot trial of cabergoline, hydergine and levodopa/carbidopa: Los Angeles Cocaine Rapid Efficacy Screening Trial (CREST). Addiction. 2005 Mar;100 Suppl 1:78-90. doi: 10.1111/j.1360-0443.2005.00991.x. PMID 15730352
- [Background] Li L, Wu Z, Cao X, Zhang L. Provider-Client Interaction in Methadone Treatment Clinics in China. J Drug Issues. 2012 Apr 1;42(2):10.1177/0022042612446593. doi: 10.1177/0022042612446593. PMID 24244048
- [Background] Li L, Liang LJ, Lin C, Feng N, Cao W, Wu Z. An intervention to improve provider-patient interaction at methadone maintenance treatment in China. J Subst Abuse Treat. 2019 Apr;99:149-155. doi: 10.1016/j.jsat.2019.01.022. Epub 2019 Feb 3. PMID 30797387
- [Background] Li L, Luo S, Lan CW, Lin C, Tuan LA, Feng N, Tuan NA. Alcohol Use, HIV Treatment Adherence, and Sexual Risk Among People with a History of Injecting Drug Use in Vietnam. AIDS Behav. 2017 Nov;21(Suppl 2):167-173. doi: 10.1007/s10461-017-1860-0. PMID 28726041
- [Background] Li L, Tuan NA, Liang LJ, Lin C, Farmer SC, Flore M. Mental health and family relations among people who inject drugs and their family members in Vietnam. Int J Drug Policy. 2013 Nov;24(6):545-9. doi: 10.1016/j.drugpo.2013.06.007. Epub 2013 Aug 1. PMID 23910167
- [Background] Li L, Hien NT, Lin C, Tuan NA, Tuan le A, Farmer SC, Detels R. An intervention to improve mental health and family well-being of injecting drug users and family members in Vietnam. Psychol Addict Behav. 2014 Jun;28(2):607-13. doi: 10.1037/a0033926. Epub 2013 Sep 30. PMID 24079647
- [Background] Holloway IW, Tan D, Gildner JL, Beougher SC, Pulsipher C, Montoya JA, Plant A, Leibowitz A. Facilitators and Barriers to Pre-Exposure Prophylaxis Willingness Among Young Men Who Have Sex with Men Who Use Geosocial Networking Applications in California. AIDS Patient Care STDS. 2017 Dec;31(12):517-527. doi: 10.1089/apc.2017.0082. PMID 29211513
- [Background] Landovitz RJ, Desmond KA, Gildner JL, Leibowitz AA. Quality of Care for HIV/AIDS and for Primary Prevention by HIV Specialists and Nonspecialists. AIDS Patient Care STDS. 2016 Sep;30(9):395-408. doi: 10.1089/apc.2016.0170. PMID 27610461
- [Background] Khuong LQ, Vu TT, Huynh VN, Thai TT. Psychometric properties of the medical outcomes study: social support survey among methadone maintenance patients in Ho Chi Minh City, Vietnam: a validation study. Subst Abuse Treat Prev Policy. 2018 Feb 14;13(1):8. doi: 10.1186/s13011-018-0147-4. PMID 29444687
- [Background] Thai TT, Jones MK, Harris LM, Heard RC. Prevalence and Correlates of Probable HIV-Associated Dementia in HIV Outpatients in Ho Chi Minh City, Vietnam. J Int Assoc Provid AIDS Care. 2017 Jul/Aug;16(4):366-375. doi: 10.1177/2325957417701195. Epub 2017 Apr 3. PMID 28367733
- [Background] Thai TT, Jones MK, Harris LM, Heard RC, Hills NK, Lindan CP. Symptoms of Depression in People Living with HIV in Ho Chi Minh City, Vietnam: Prevalence and Associated Factors. AIDS Behav. 2018 Jul;22(Suppl 1):76-84. doi: 10.1007/s10461-017-1946-8. PMID 29079945
- [Background] Thai TT, Jones MK, Harris LM, Heard RC. The association between symptoms of mental disorders and health risk behaviours in Vietnamese HIV positive outpatients: a cross-sectional study. BMC Public Health. 2017 Mar 14;17(1):250. doi: 10.1186/s12889-017-4162-6. PMID 28288615
- [Background] Schmidt LG, Siemetzki H. [A differential effect profile of neuroleptic therapy of acute schizophrenic patients? Results of a clinico-naturalistic study]. Nervenarzt. 1988 Dec;59(12):721-6. No abstract available. German. PMID 2905770
- [Background] Shoptaw S, Landovitz RJ, Reback CJ. Contingent Vs. Non-Contingent Rewards: Time-Based Intervention Response Patterns Among Stimulant-Using Men Who Have Sex With Men. J Subst Abuse Treat. 2017 Jan;72:19-24. doi: 10.1016/j.jsat.2016.09.004. Epub 2016 Sep 13. PMID 27938777
- [Background] Shoptaw S, Reback CJ, Peck JA, Yang X, Rotheram-Fuller E, Larkins S, Veniegas RC, Freese TE, Hucks-Ortiz C. Behavioral treatment approaches for methamphetamine dependence and HIV-related sexual risk behaviors among urban gay and bisexual men. Drug Alcohol Depend. 2005 May 9;78(2):125-34. doi: 10.1016/j.drugalcdep.2004.10.004. Epub 2004 Nov 28. PMID 15845315
- [Background] Shoptaw S, Reback CJ, Larkins S, Wang PC, Rotheram-Fuller E, Dang J, Yang X. Outcomes using two tailored behavioral treatments for substance abuse in urban gay and bisexual men. J Subst Abuse Treat. 2008 Oct;35(3):285-93. doi: 10.1016/j.jsat.2007.11.004. Epub 2008 Mar 7. PMID 18329226
- [Background] Landovitz RJ, Fletcher JB, Inzhakova G, Lake JE, Shoptaw S, Reback CJ. A novel combination HIV prevention strategy: post-exposure prophylaxis with contingency management for substance abuse treatment among methamphetamine-using men who have sex with men. AIDS Patient Care STDS. 2012 Jun;26(6):320-8. doi: 10.1089/apc.2011.0432. PMID 22680280
- [Background] Landovitz RJ, Fletcher JB, Shoptaw S, Reback CJ. Contingency management facilitates the use of postexposure prophylaxis among stimulant-using men who have sex with men. Open Forum Infect Dis. 2015 Jan 1;2(1):ofu114. doi: 10.1093/ofid/ofu114. eCollection 2015 Jan. PMID 25884003
- [Background] Reback CJ, Shoptaw S. Development of an evidence-based, gay-specific cognitive behavioral therapy intervention for methamphetamine-abusing gay and bisexual men. Addict Behav. 2014 Aug;39(8):1286-91. doi: 10.1016/j.addbeh.2011.11.029. Epub 2011 Nov 26. PMID 22169619
- [Background] Reback CJ, Veniegas R, Shoptaw S. Getting Off: development of a model program for gay and bisexual male methamphetamine users. J Homosex. 2014;61(4):540-53. doi: 10.1080/00918369.2014.865459. PMID 24245506
- [Background] Shoptaw S, Reback C, Peck JA, Larkins S, Freese TE, Rawson RA. Getting Off: A Behavioral Treatment Intervention for Gay and Bisexual Methamphetamine Users [Internet]. 2005 [cited 2017 Mar 31]. Available from: http://friendscommunitycenter.org/documents/Getting_Off_Treatment_Manual.pdf
- [Background] Reback CJ, Shoptaw S, Riley J, Stone K. Getting Off: A Behavioral Treatment Intervention for Gay and Bisexual Methamphetamine Users. A Training Manual for Counselors [Internet]. 2008 [cited 2017 Mar 31]. Available from: http://friendscommunitycenter.org/documents/Getting_Off_Counselor_Training_Manual.pdf
- [Background] Collins LM, Murphy SA, Bierman KL. A conceptual framework for adaptive preventive interventions. Prev Sci. 2004 Sep;5(3):185-96. doi: 10.1023/b:prev.0000037641.26017.00. PMID 15470938
- [Background] Rees RJ. Leprosy. A preliminary review of the experimental evaluation of drugs for the treatment of leprosy. Trans R Soc Trop Med Hyg. 1967;61(4):581-95. doi: 10.1016/0035-9203(67)90111-3. No abstract available. PMID 4167891
- [Background] Lei H, Nahum-Shani I, Lynch K, Oslin D, Murphy SA. A "SMART" design for building individualized treatment sequences. Annu Rev Clin Psychol. 2012;8:21-48. doi: 10.1146/annurev-clinpsy-032511-143152. Epub 2011 Dec 12. PMID 22224838
- [Background] Belzer ME, MacDonell KK, Ghosh S, Naar S, McAvoy-Banerjea J, Gurung S, Cain D, Fan CA, Parsons JT. Adaptive Antiretroviral Therapy Adherence Interventions for Youth Living With HIV Through Text Message and Cell Phone Support With and Without Incentives: Protocol for a Sequential Multiple Assignment Randomized Trial (SMART). JMIR Res Protoc. 2018 Dec 20;7(12):e11183. doi: 10.2196/11183. PMID 30573448
- [Background] Mimiaga MJ, Kuhns LM, Biello KB, Olson J, Hoehnle S, Santostefano CM, Hughto JMW, Safi H, Salhaney P, Chen D, Garofalo R. Positive STEPS - a randomized controlled efficacy trial of an adaptive intervention for strengthening adherence to antiretroviral HIV treatment among youth: study protocol. BMC Public Health. 2018 Jul 13;18(1):867. doi: 10.1186/s12889-018-5815-9. PMID 30001703
- [Background] Grant S, Agniel D, Almirall D, Burkhart Q, Hunter SB, McCaffrey DF, Pedersen ER, Ramchand R, Griffin BA. Developing adaptive interventions for adolescent substance use treatment settings: protocol of an observational, mixed-methods project. Addict Sci Clin Pract. 2017 Dec 19;12(1):35. doi: 10.1186/s13722-017-0099-4. PMID 29254500
- [Background] Apostolopoulos Y, Lemke MK, Barry AE, Lich KH. Moving alcohol prevention research forward-Part I: introducing a complex systems paradigm. Addiction. 2018 Feb;113(2):353-362. doi: 10.1111/add.13955. Epub 2017 Aug 25. PMID 28734094
- [Background] Bortolon CB, Moreira TC, Signor L, Guahyba BL, Figueiro LR, Ferigolo M, Barros HM. Six-Month Outcomes of a Randomized, Motivational Tele-intervention for Change in the Codependent Behavior of Family Members of Drug Users. Subst Use Misuse. 2017 Jan 28;52(2):164-174. doi: 10.1080/10826084.2016.1223134. Epub 2016 Oct 18. PMID 27754731
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Damschroder LJ, Hagedorn HJ. A guiding framework and approach for implementation research in substance use disorders treatment. Psychol Addict Behav. 2011 Jun;25(2):194-205. doi: 10.1037/a0022284. PMID 21443291
- [Background] Green HD. A Community-Based Evaluation of Screening, Brief Intervention, and Referral to Treatment (SBIRT) for the Black Community. Qual Health Res. 2018 Feb;28(3):418-432. doi: 10.1177/1049732317746962. Epub 2017 Dec 18. PMID 29254450
- [Background] Sorensen JL, Kosten T. Developing the tools of implementation science in substance use disorders treatment: applications of the consolidated framework for implementation research. Psychol Addict Behav. 2011 Jun;25(2):262-8. doi: 10.1037/a0022765. PMID 21668086
- [Background] VanDevanter N, Kumar P, Nguyen N, Nguyen L, Nguyen T, Stillman F, Weiner B, Shelley D. Application of the Consolidated Framework for Implementation Research to assess factors that may influence implementation of tobacco use treatment guidelines in the Viet Nam public health care delivery system. Implement Sci. 2017 Feb 28;12(1):27. doi: 10.1186/s13012-017-0558-z. PMID 28241770
- [Background] Pollack TM, Duong HT, Pham TT, Nguyen TD, Libman H, Ngo L, McMahon JH, Elliott JH, Do CD, Colby DJ. Routine versus Targeted Viral Load Strategy among Patients Starting Antiretroviral in Hanoi, Vietnam. J Int AIDS Soc. 2019 Mar;22(3):e25258. doi: 10.1002/jia2.25258. PMID 30897303
- [Background] Wingood GM, DiClemente RJ. The ADAPT-ITT model: a novel method of adapting evidence-based HIV Interventions. J Acquir Immune Defic Syndr. 2008 Mar 1;47 Suppl 1:S40-6. doi: 10.1097/QAI.0b013e3181605df1. PMID 18301133
- [Background] Khumsaen N, Stephenson R. Adaptation of the HIV/AIDS Self-Management Education Program for Men Who Have Sex With Men in Thailand: An Application of the ADAPT-ITT Framework. AIDS Educ Prev. 2017 Oct;29(5):401-417. doi: 10.1521/aeap.2017.29.5.401. PMID 29068714
- [Background] Muhr T. Atlas.ti. Berlin: Scientific Software Development; 1997.
- [Background] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Miller WR, Tonigan JS. Assessing drinkers' motivation for change: The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES). Psychol Addict Behav. 19960101;10(2):81.
- [Background] McLellan AT, Kushner H, Metzger D, Peters R, Smith I, Grissom G, Pettinati H, Argeriou M. The Fifth Edition of the Addiction Severity Index. J Subst Abuse Treat. 1992;9(3):199-213. doi: 10.1016/0740-5472(92)90062-s. PMID 1334156
- [Background] Martin GW, Wilkinson DA, Poulos CX. The Drug Avoidance Self-Efficacy Scale. J Subst Abuse. 1995;7(2):151-63. doi: 10.1016/0899-3289(95)90001-2. PMID 7580226
- [Background] Twitchell GR, Huber A, Reback CJ, Shoptaw S. Comparison of General and Detailed HIV Risk Assessments Among Methamphetamine Abusers. AIDS Behav. 2002 Jun 1;6(2):153-162.
- [Background] McGregor C, Srisurapanont M, Mitchell A, Longo MC, Cahill S, White JM. Psychometric evaluation of the Amphetamine Cessation Symptom Assessment. J Subst Abuse Treat. 2008 Jun;34(4):443-9. doi: 10.1016/j.jsat.2007.05.007. Epub 2007 Jul 13. PMID 17629443
- [Background] DiIorio C, Maibach E, O'Leary A, Sanderson CA, Celentano D. Measurement of condom use self-efficacy and outcome expectancies in a geographically diverse group of STD patients. AIDS Educ Prev. 1997 Feb;9(1):1-13. PMID 9083587
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Chesney MA, Ickovics JR, Chambers DB, Gifford AL, Neidig J, Zwickl B, Wu AW. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committee of the Adult AIDS Clinical Trials Group (AACTG). AIDS Care. 2000 Jun;12(3):255-66. doi: 10.1080/09540120050042891. PMID 10928201
- [Background] NIDA. Seek, Test, Treat and Retain: Addressing HIV among Vulnerable Populations [Internet]. 2013 [cited 2018 Nov 15]. Available from: https://www.drugabuse.gov/researchers/research-resources/data-harmonization-projects/seek-test-treat-retain/addressing-hiv-among-vulnerable-populations
- [Background] ZUNG WW. A SELF-RATING DEPRESSION SCALE. Arch Gen Psychiatry. 1965 Jan;12:63-70. doi: 10.1001/archpsyc.1965.01720310065008. No abstract available. PMID 14221692
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Sarason IG, Levine HM, Basham RB, Sarason BR. Assessing social support: The social support questionnaire. J Pers Soc Psychol. 1983;139.
- [Background] Willer B, Ottenbacher KJ, Coad ML. The community integration questionnaire. A comparative examination. Am J Phys Med Rehabil. 1994 Apr;73(2):103-11. doi: 10.1097/00002060-199404000-00006. PMID 8148099
- [Background] Stambaugh D. Holding rabbits. J Biol Photogr. 1987 Jul;55(3):77. No abstract available. PMID 3680138
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Vuong T, Ritter A, Shanahan M, Ali R, Nguyen N, Pham K, Vuong TTA, Le GM. Outcomes of compulsory detention compared to community-based voluntary methadone maintenance treatment in Vietnam. J Subst Abuse Treat. 2018 Apr;87:9-15. doi: 10.1016/j.jsat.2018.01.011. Epub 2018 Jan 16. PMID 29471930
- [Background] UNAIDS. Costing Guidelines for HIV Prevention Strategies. UNAIDS (Geneva); 2000 p. 140.
- [Background] Shoptaw S, Klausner JD, Reback CJ, Tierney S, Stansell J, Hare CB, Gibson S, Siever M, King WD, Kao U, Dang J. A public health response to the methamphetamine epidemic: the implementation of contingency management to treat methamphetamine dependence. BMC Public Health. 2006 Aug 18;6:214. doi: 10.1186/1471-2458-6-214. PMID 16919170
- [Background] Hintz J. PASS 12. Kaysville, Utah, USA: NCSS, LLC www.ncss.com; 2013.
- [Background] Nahum-Shani I, Qian M, Almirall D, Pelham WE, Gnagy B, Fabiano GA, Waxmonsky JG, Yu J, Murphy SA. Experimental design and primary data analysis methods for comparing adaptive interventions. Psychol Methods. 2012 Dec;17(4):457-477. doi: 10.1037/a0029372. Epub 2012 Oct 1. PMID 23025433
- [Background] Neumann PJ, Sanders GD, Russell LB, Siegel JE, Ganiats TG, editors. Cost effectiveness in health and medicine. Second edition. Oxford ; New York: Oxford University Press; 2017.
- [Background] Creswell JW. Designing and conducting mixed methods research. 2nd ed. Los Angeles: SAGE Publications; 2011
- [Background] Bui HTM, Le GM, Mai AQ, Zablotska-Manos I, Maher L. Barriers to access and uptake of antiretroviral therapy among HIV-positive men who have sex with men in Hanoi, Vietnam: from HIV testing to treatment. Cult Health Sex. 2017 Aug;19(8):859-872. doi: 10.1080/13691058.2016.1269203. Epub 2017 Jan 19. PMID 28100136
- [Background] Itakura T, Okuno T, Ueno M, Nakakita K, Nakai K, Naka Y, Imai H, Kamei I, Komai N. Immunohistochemical demonstration of vasopressin nerve fibers in the cerebral artery. J Cereb Blood Flow Metab. 1988 Aug;8(4):606-8. doi: 10.1038/jcbfm.1988.102. PMID 3392119
- [Background] Vuong T, Nguyen N, Le G, Shanahan M, Ali R, Ritter A. The political and scientific challenges in evaluating compulsory drug treatment centers in Southeast Asia. Harm Reduct J. 2017 Jan 11;14(1):2. doi: 10.1186/s12954-016-0130-1. PMID 28077147
- [Background] Hoang TV, Ha TT, Hoang TM, Nhu NT, Quoc NC, Tam Nt, Mills S. Impact of a methadone maintenance therapy pilot in Vietnam and its role in a scaled-up response. Harm Reduct J. 2015 Oct 16;12:39. doi: 10.1186/s12954-015-0075-9. PMID 26471235
- [Derived] Diep NB, Trang NT, Huy DD, Van HTH, Truc TT, Van Dung D, Li MJ, Shoptaw SJ, Li L, Giang LM. Non-adherence to treatment and concurrent opioid use among people on methadone maintenance treatment using methamphetamine in Vietnam. J Subst Use Addict Treat. 2025 Jun;173:209686. doi: 10.1016/j.josat.2025.209686. Epub 2025 Mar 27. PMID 40157650
- [Derived] Giang LM, Trang NT, Thuy DT, Nguyen HH, Diep NB, Van HTH, Truc TT, Reback CJ, Li M, Van Dung D, Shoptaw S. Using ADAPT-ITT framework to tailor evidence-based interventions for addressing methamphetamine use among methadone patients in Vietnam. Drug Alcohol Rev. 2023 Nov;42(7):1667-1679. doi: 10.1111/dar.13739. Epub 2023 Aug 23. PMID 37614129
- [Derived] Giang LM, Trang NT, Diep NB, Thuy DTD, Thuy DT, Hoe HD, Van HTH, Truc TT, Nguyen HH, Lai NL, Linh PTD, Vi VTT, Reback CJ, Leibowitz A, Li L, Lin C, Li M, Do Van Dung, Shoptaw S. An adaptive design to screen, treat, and retain people with opioid use disorders who use methamphetamine in methadone clinics (STAR-OM): study protocol of a clinical trial. Trials. 2022 Apr 23;23(1):342. doi: 10.1186/s13063-022-06278-w. PMID 35461300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began on 29 June 2021 and ended 1 April 2023. We screened 6708 people with opioid use disorder from 15 methadone clinics in Hanoi and Ho Chi Minh City and enrolled 667 participants.
Pre-assignment Details: After enrollment, 2 participants withdrew consent and declined to participate in the intervention. Thus, they were not randomized.
  This study employed a Sequential Multiple Assignment Randomized Trial (SMART) design. In the first phase, participants were randomized to one of two frontline interventions for 12 weeks. At Week 13, they were re-assigned to one of three adaptive strategies for an additional 12 weeks. We report outcomes stratified by the initial frontline intervention groups.
Groups:
- High Intensity Frontline Intervention: Participants randomized to the high intensity frontline intervention arm (12 weeks of contingency management)
- Low Intensity Frontline Intervention: Participants randomized into the low intensity frontline intervention arm (6 weeks of contingency management plus 6 weeks of group education)
- Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2: The high-intensity frontline intervention consisted of 12 weeks of Contingency Management (CM), delivered through rewards for methamphetamine-negative urine samples. Participants who responded to Stage 1 continued to receive SMS reminders in Stage 2. SMS consisted of two daily reminders plus one weekly self-monitoring assessment, delivered for 12 weeks. This intervention was a Stage 2 add-on intervention for Stage 1 responders.
- Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2: The high-intensity frontline intervention consisted of 12 weeks of CM. Participants who did not respond to Stage 1 were randomized and received the Matrix intervention in Stage 2, attending 12 weekly group counseling sessions. This intervention was a Stage 2 add-on intervention for Stage 1 non-responders.
- Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2: The high-intensity frontline intervention consisted of 12 weeks of CM. Participants who did not respond to Stage 1 were randomized and received the Matrix + CM intervention in Stage 2, attending 12 weekly Matrix group counseling sessions plus 12 weeks of CM. This intervention was a Stage 2 add-on intervention for Stage 1 non-responders.
- Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2: The low-intensity frontline intervention consisted of 6 weeks of CM, followed by 6 weeks of Group Education (GE). Participants who responded to Stage 1 continued to receive SMS reminders in Stage 2, consisting of two daily reminders plus one weekly self-monitoring assessment delivered for 12 weeks. This intervention was a Stage 2 add-on intervention for Stage 1 responders.
- Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2: The low-intensity frontline intervention consisted of 6 weeks of CM, followed by 6 weeks of GE. Participants who did not respond to Stage 1 were randomized and received the Matrix intervention in Stage 2, attending 12 weekly group counseling sessions. This intervention was a Stage 2 add-on intervention for Stage 1 non-responders.
- Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2: The low-intensity frontline intervention consisted of 6 weeks of CM, followed by 6 weeks of GE. Participants who did not respond to Stage 1 were randomized and received the Matrix + CM intervention in Stage 2, attending 12 weekly Matrix group counseling sessions plus 12 weeks of CM. This intervention was a Stage 2 add-on intervention for Stage 1 non-responders.
Period: Stage 1 Intervention (Weeks 0 to 12)
Arm/Group | High Intensity Frontline Intervention | Low Intensity Frontline Intervention | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Started | 328 | 337 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 315 | 328 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 Intervention (Weeks 13 to 26)
Arm/Group | High Intensity Frontline Intervention | Low Intensity Frontline Intervention | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Started | 0 | 0 | 230 | 40 | 45 | 198 | 68 | 62
Completed | 0 | 0 | 220 | 30 | 41 | 189 | 64 | 55
Not Completed | 0 | 0 | 10 | 10 | 4 | 9 | 4 | 7

BASELINE CHARACTERISTICS:
Population: During the frontline intervention stage (Weeks 1-12), participants were randomized into two groups. Therefore, we analyzed baseline data according to these two groups. In the second phase, participants were re-assigned to one of three adaptive intervention groups based on their response in the first phase, with each original group branching into all three adaptive arms.
Groups:
- High Intensity Frontline Intervention: Participants randomized to the high intensity frontline intervention (12 weeks of contingency management)
- Low Intensity Frontline Intervention: Participants randomized to the low intensity frontline intervention (6 weeks of contingency management plus 6 weeks of group education)
- Total: Total of all reporting groups
Arm/Group | High Intensity Frontline Intervention | Low Intensity Frontline Intervention | Total
Number analyzed (Participants) | 328 | 337 | 665
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (7.2) | 41.5 (7.5) | 41.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 35 | 39 | 74
    Male | 293 | 298 | 591
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 328 | 337 | 665
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 328 | 337 | 665
Alcohol, Smoking and Substance Involvement Screening Test [Mean (Standard Deviation); unit: units on a scale] — The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) detects problematic substance use. The tool consists of 8 core questions for each substance assessing lifetime use, use in the past 3 months and problems related to use. Each substance receives a score ranging from 0 to 39. For alcohol, the cut-off threshold for Low risk is 0-10, for Moderate risk is 11-26 and for High risk is 27+. For other substance, the cut-off threshold for Low risk is 0-3, for Moderate risk is 4 to 26 and for High risk is 27+.
  In this study, we only use ASSIST for methamphetamine.
  units on a scale | 16.3 (8.1) | 16.7 (8.3) | 16.5 (8.2)
HIV status [Count of Participants; unit: Participants] — Quick screening test - Participants who screened positive received a subsequent confirmatory HIV test.
  Participants
    Negative | 271 | 262 | 533
    Positive | 57 | 75 | 132
Currently married [Count of Participants; unit: Participants]
  No | 179 | 198 | 377
  Yes | 149 | 139 | 288
Education [Count of Participants; unit: Participants]
  Less than 12th grade | 225 | 242 | 467
  12th grade or higher | 103 | 95 | 198
Has a paid job [Count of Participants; unit: Participants]
  No | 125 | 124 | 249
  Yes | 203 | 213 | 416
Methamphetamine urine drug screen [Count of Participants; unit: Participants]
  Negative | 130 | 122 | 252
  Positive | 198 | 215 | 413

OUTCOME MEASURES:

1. Primary Outcome: Increase in HIV Viral Suppression for HIV-positive Participants: High- vs. Low-Intensity Frontline Intervention With SMS in Stage 2
Description: HIV viral load was assessed at baseline (Week 0), Week 13, and Week 24 after enrollment. Viral load was categorized as: ≥200 copies/mL; ≥20 to <200 copies/mL; or undetectable (<20 copies/mL). This outcome measure reports viral suppression status at baseline (Week 0) and Week 24 in order to evaluate change in viral suppression following completion of the full intervention period.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 responders with completed viral load assessments at week 24 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2
Number analyzed (Participants) | 40 | 43
Participants
  Baseline: Undetected or <20copies/mL | 31 | 35
  Baseline: >=20 copies/mL & <200 copies/mL | 6 | 3
  Baseline: >= 200 copies/mL | 3 | 5
  Week 24: Undetected or <20copies/mL | 33 | 39
  Week 24: >=20 copies/mL & <200 copies/mL | 3 | 1
  Week 24: >= 200 copies/mL | 4 | 3
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Baseline comparison; Test type: Superiority; p = 0.447, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison; Test type: Superiority; p = 0.491, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05

2. Primary Outcome: Increase in HIV Viral Suppression for HIV-positive Participants: High- vs. Low-Intensity Frontline Intervention With Matrix/Matrix + CM in Stage 2
Description: HIV viral load was assessed at baseline (Week 0), Week 13, and Week 24 after enrollment. Viral load was categorized as: ≥200 copies/mL; ≥20 to <200 copies/mL; or undetectable (<20 copies/mL). This outcome measure reports viral suppression status at baseline (Week 0) and Week 24 in order to evaluate the change in viral suppression following completion of the full intervention period.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 non-responders with completed viral load assessments at week 24 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Number analyzed (Participants) | 6 | 11 | 6 | 12
Participants
  Baseline: Undetected or < 20 copies/mL | 4 | 10 | 6 | 8
  Baseline: ≥ 20 copies/mL & < 200 copies/mL | 1 | 0 | 0 | 1
  Baseline: ≥ 200 copies/mL | 1 | 1 | 0 | 3
  Week 24: Undetected or < 20 copies/mL | 5 | 9 | 4 | 9
  Week 24: ≥ 20 copies/mL & < 200 copies/mL | 1 | 0 | 1 | 0
  Week 24: ≥ 200 copies/mL | 0 | 2 | 1 | 3
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Baseline comparison; Test type: Superiority; p = 0.600, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison; Test type: Superiority; p = 0.495, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05

3. Primary Outcome: Reduction in HIV Risk Behaviors for Both HIV-positive and HIV-negative Participants: High- vs. Low-Intensity Frontline Intervention With SMS in Stage 2
Description: Structured questionnaires will collect self-reported data at baseline and week 24 after enrolment.
  HIV risk behaviors were grouped into two types:
  1. sexual risk behaviors, such as having sex with partners who were HIV-positive or whose status was unknown, having sex while using drugs or alcohol, or using methamphetamine to find partners or enhance sex
  2. needle/syringe risk behaviors, such as reusing needles or syringes that had already been used by others (even if cleaned) or reusing their own needles or syringes multiple times.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 responders with completed assessments at week 24 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2
Number analyzed (Participants) | 222 | 192
Participants
  Baseline: Sexual risk behaviors: Yes | 41 | 24
  Baseline: Sexual risk behaviors: No | 181 | 168
  Week 24: Sexual risk behaviors: Yes | 16 | 14
  Week 24: Sexual risk behaviors: No | 206 | 178
  Baseline: HIV needle/syringe risk behaviors: Yes | 0 | 3
  Baseline: HIV needle/syringe risk behaviors: No | 222 | 189
  Week 24: HIV needle/syringe risk behaviors: Yes | 0 | 1
  Week 24: HIV needle/syringe risk behaviors: No | 222 | 191
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Baseline comparison regarding sexual risk behaviors; Test type: Superiority; p = 0.096, Chi-squared — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Baseline comparison regarding HIV needle/syringe risk behaviors; Test type: Superiority; p = 0.098, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 3: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison regarding sexual risk behaviors; Test type: Superiority; p = 0.974, Chi-squared — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 4: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison regarding HIV needle/syringe risk behaviors; Test type: Superiority; p = 0.464, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05

4. Primary Outcome: Reduction in HIV Risk Behaviors for Both HIV-positive and HIV-negative Participants: High- vs. Low-Intensity Frontline Intervention With Matrix/Matrix + CM in Stage 2
Description: Structured questionnaires will collect self-reported data at baseline and 24 weeks after enrolment.
  HIV risk behaviors were grouped into two types:
  1. sexual risk behaviors, such as having sex with partners who were HIV-positive or whose status was unknown, having sex while using drugs or alcohol, or using methamphetamine to find partners or enhance sex.
  2. needle/syringe risk behaviors, such as reusing needles or syringes that had already been used by others (even if cleaned) or reusing their own needles or syringes multiple times.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 non-responders with completed assessments at week 24 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Number analyzed (Participants) | 33 | 65 | 41 | 56
Participants
  Baseline: Sexual risk behaviors: Yes | 5 | 13 | 8 | 13
  Baseline: Sexual risk behaviors: No | 28 | 52 | 33 | 43
  Week 24: Sexual risk behaviors: Yes | 3 | 8 | 4 | 10
  Week 24: Sexual risk behaviors: No | 30 | 57 | 37 | 46
  Baseline: HIV needle/syringe risk behaviors: Yes | 0 | 1 | 0 | 1
  Baseline: HIV needle/syringe risk behaviors: No | 33 | 64 | 41 | 55
  Week 24: HIV needle/syringe risk behaviors: Yes | 0 | 0 | 2 | 0
  Week 24: HIV needle/syringe risk behaviors: No | 33 | 65 | 39 | 56
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Baseline comparison regarding sexual risk behaviors; Test type: Superiority; p = 0.835, Chi-squared — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison regarding sexual risk behaviors; Test type: Superiority; p = 0.610, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 3: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Baseline comparison regarding HIV needle/syringe risk behaviors; Test type: Superiority; p = 1.000, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05
Statistical Analysis 4: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison regarding HIV needle/syringe risk behaviors; Test type: Superiority; p = 0.071, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05

5. Secondary Outcome: Heroin-negative Test: High- vs. Low-Intensity Frontline Intervention
Description: Heroin use was measured using twice-weekly urine drug tests. Participants were classified as heroin-negative if all four urine drug tests conducted during Weeks 11-12 and during Weeks 24-25 were negative for heroin.
Time Frame: Weeks 11-12 (end of Stage 1) and Weeks 24-25 (end of Stage 2)
Population: Participants were analyzed according to their Stage 1 intervention assignment. Although participants could be re-randomized to different intervention groups in Stage 2, Stage 2 assignments were not considered in this analysis. Heroin-negative after Stage 2 was compared based on participants' original Stage 1 group.
Measure: Count of Participants; unit: Participants
Groups:
- Received High Intensity Frontline Intervention in Stage 1: The high-intensity frontline intervention consisted of 12 weeks of contingency management in Stage 1, delivered through rewards for methamphetamine-negative urine samples.
- Received Low Intensity Frontline Intervention in Stage 1: The low-intensity frontline intervention consisted of 6 weeks of contingency management followed by 6 weeks of group education in Stage 1.
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 | Received Low Intensity Frontline Intervention in Stage 1
Number analyzed (Participants) | 328 | 337
Participants
  Week 12 | 252 | 237
  Week 25 | 238 | 248
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 vs Received Low Intensity Frontline Intervention in Stage 1; Week 12 comparison; Test type: Superiority; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.08 to 2.61]
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 vs Received Low Intensity Frontline Intervention in Stage 1; Week 25 comparison; Test type: Superiority; p = 0.404, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.76 to 2.01]

6. Secondary Outcome: Heroin-negative Test: Matrix vs. Matrix + CM Adaptive Intervention
Description: Heroin use was measured using twice-weekly urine drug tests. Participants were classified as heroin-negative if all four urine drug tests conducted during Weeks 24-25 were negative for heroin.
Time Frame: Week 24-25 (end of Stage 2)
Population: Heroin -negative among non-responders who were re-randomized to the Matrix intervention in Stage 2 are compared to non-responders who were re-randomized to the Matrix + contingency management in Stage 2; data are aggregated over both Stage 1 interventions.
Measure: Count of Participants; unit: Participants
Groups:
- Received Matrix in Stage 2: Participants who did not have a response in Stage 1 and were re-randomized to the Matrix intervention in Stage 2 attended 12 weekly group counseling sessions.
- Received Matrix + Contingency Management in Stage 2: Participants who did not have a response in Stage 1 and were re-randomized to the Matrix + contingency management in Stage 2 attended 12 weekly Matrix group counseling sessions plus 12 weeks of contingency management delivered twice weekly.
Arm/Group | Received Matrix in Stage 2 | Received Matrix + Contingency Management in Stage 2
Number analyzed (Participants) | 108 | 107
Participants | 48 | 50
Statistical Analysis 1: Comparison: Received Matrix in Stage 2 vs Received Matrix + Contingency Management in Stage 2; Test type: Superiority; p = 0.737, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.53 to 1.56]

7. Secondary Outcome: Adherence to ART if HIV-positive: High- vs. Low-Intensity Frontline Intervention With SMS in Stage 2
Description: This information will be collected using the study questionnaire at baseline, weeks 12th, and 24th.
  People who adhered to ART was defined as currently on ART and either (1) within 4 days they never forgot to take HIV medication or (2) never took HIV medication later 2 hours than required or (3) forgot to take their HIV medication at the weekend. This outcome measure reports ART adherence at baseline (Week 0) and Week 24 in order to evaluate change in ART adherence following completion of the full intervention period.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 responders who completed the Week 24 assessment and received ART were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2
Number analyzed (Participants) | 38 | 41
Participants
  Baseline: Adherence to ART | 38 | 41
  Baseline: Non-adherence to ART | 0 | 0
  Week 24: Adherence to ART | 37 | 37
  Week 24: Non-adherence to ART | 1 | 4
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 25 comparison; No test for baseline due to all adhering to ART; Test type: Superiority; p = 0.361, Fisher Exact — The threshold for statistical significance for all analyses was set to p = 0.05

8. Secondary Outcome: Adherence to ART if HIV-positive: High- vs. Low-Intensity Frontline Intervention With Matrix/Matrix + CM in Stage 2
Description: This information will be collected using the study questionnaire at baseline, weeks 12th and 24th.
  People who adhered to ART was defined as currently on ART and either (1) within 4 days they never forgot to take HIV medication or (2) never took HIV medication later 2 hours than required or (3) forgot to take their HIV medication at the weekend. This outcome measure reports ART adherence at baseline (Week 0) and Week 24 in order to evaluate change in ART adherence following completion of the full intervention period.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 non-responders who completed the Week 24 assessment and received ART were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Number analyzed (Participants) | 7 | 12 | 6 | 12
Participants
  Baseline: Adherence to ART | 6 | 12 | 6 | 10
  Baseline: Non-adherence to ART | 1 | 0 | 0 | 0
  Baseline: HIV seroconversion by Week 24 / ART discontinuation by Week 24 | 0 | 0 | 0 | 2
  Week 24: Adherence to ART | 7 | 11 | 6 | 12
  Week 24: Non-adherence to ART | 0 | 0 | 0 | 0
  Week 24: HIV seroconversion by Week 24 / ART discontinuation by Week 24 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Baseline comparison; Test type: Superiority; p = 0.371, Fisher Exact

9. Secondary Outcome: Frequency of HIV Testing if HIV-negative: High- vs. Low-Intensity Frontline Intervention With SMS in Stage 2
Description: HIV testing will be assessed based on whether HIV-negative participants received HIV testing services at each assessment point
Time Frame: Week 12 (end of Stage 1) and Week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 responders with completed assessments at week 12 and week 24 and HIV-negative were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2
Number analyzed (Participants) | 181 | 149
Participants
  Week 12 | 181 | 148
  Week 24 | 179 | 149
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 12 comparison of groups on HIV testing; Test type: Superiority; p = 0.451, Fisher Exact
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison of groups on HIV testing; Test type: Superiority; p = 0.503, Fisher Exact

10. Secondary Outcome: Frequency of HIV Testing if HIV-negative: High- vs. Low-Intensity Frontline Intervention With Matrix/Matrix + CM in Stage 2
Description: as for outcome 9
Time Frame: Week 12 (end of Stage 1) and Week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 non-responders with completed assessments at week 12 and week 24 and HIV-negative were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Number analyzed (Participants) | 26 | 52 | 35 | 44
Participants
  Week 12 | 25 | 52 | 35 | 43
  Week 24 | 26 | 52 | 35 | 44
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 12 comparison of groups on HIV testing; Test type: Superiority; p = 0.320, Fisher Exact
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison of groups on HIV testing; Test type: Superiority; p = 1.000, Fisher Exact; All HIV-negative participants received HIV testing; therefore, no variability exists between groups for statistical comparison

11. Secondary Outcome: Frequency of Opioid Overdose: High- vs. Low-Intensity Frontline Intervention With SMS in Stage 2
Description: Opioid overdose will be assessed in the past 3 months through participant self-report using the question: "In the past 3 months, how many times have you had an opioid/heroin overdose?". Overdose is defined as an acute event due to heroin or other opioid use that required assistance from another person to recover (e.g., ambulance call, resuscitation, being awakened by others). This definition excludes episodes where the participant "just slept it off." Both non-fatal and fatal overdoses are included, and intentional overdoses (suicidal attempts) are also counted. For analysis, participants reporting at least one overdose in the past 3 months will be categorized as "Yes" for having experienced an overdose.
Time Frame: Week 12 (end of Stage 1) and Week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 responders with completed assessments at week 12 and week 24 were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2
Number analyzed (Participants) | 222 | 192
Participants
  Week 12 | 1 | 0
  Week 24 | 0 | 0
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 12 comparison of groups on opioid overdose; Test type: Superiority; p > 0.99, Fisher Exact
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison of groups on opioid overdose; Test type: Superiority; p = 1.000, Fisher Exact; No test due to zero cell counts

12. Secondary Outcome: Frequency of Opioid Overdose: High- vs. Low-Intensity Frontline Intervention With Matrix/Matrix + CM in Stage 2
Description: as for outcome 11
Time Frame: Week 12 (end of Stage 1) and Week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 non-responders with completed assessments at week 12 and week 24 were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Number analyzed (Participants) | 31 | 64 | 41 | 56
Participants
  Week 12 | 1 | 0 | 0 | 0
  Week 24 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 12 comparison of groups on opioid overdose; Test type: Superiority; p = 0.166, Fisher Exact
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison of groups on opioid overdose; Test type: Superiority; p = 1.000, Fisher Exact; No test due to zero cell counts

13. Secondary Outcome: Changes in Quality of Life: High- vs. Low-Intensity Frontline Intervention With SMS in Stage 2
Description: Quality of life will be assessed using the EQ-5D-5L instrument, which includes five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity. Responses will be converted into a single utility index score using the Vietnamese value set (https://doi.org/10.1007/s11136-020-02469-7), ranging from 0-1, where higher scores indicate better health-related quality of life. In addition, participants will rate their overall health on the EQ Visual Analogue Scale (VAS), ranging from 0 ("worst imaginable health") to 100 ("best imaginable health"), with higher scores reflecting better perceived health. Both the EQ-5D-5L utility index and the VAS score will be analyzed as continuous outcomes.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 responders with completed assessments at week 24 were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2
Number analyzed (Participants) | 222 | 192
score on a scale
  Baseline EQ-5D-5L value | 0.9 (0.1) | 0.9 (0.1)
  Baseline VAS | 74.8 (14.7) | 74.4 (14.9)
  Week 24 EQ-5D-5L value | 1.0 (0.1) | 1.0 (0.1)
  Week 24 VAS | 78.2 (12.5) | 75.9 (14.3)
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Baseline comparison of groups on quality of life value; Test type: Superiority; p = 0.280, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Baseline comparison of groups on VAS score; Test type: Superiority; p = 0.812, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison of groups on quality of life value; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Received High Intensity Frontline Intervention in Stage 1 and SMS in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and SMS in Stage 2; Week 24 comparison of groups on VAS score; Test type: Superiority; p = 0.184, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Reduction in Methamphetamine Use: High- vs. Low-Intensity Frontline Intervention
Description: Methamphetamine use was measured using twice-weekly urine drug tests. Treatment response is defined as testing methamphetamine-negative in 4 out of a possible 4 urine tests during Weeks 11-12 and during Weeks 24-25.
Time Frame: Weeks 11-12 (end of Stage 1) and week 24-25 (end of Stage 2)
Population: Participants were analyzed according to their Stage 1 intervention assignment. Although participants could be re-randomized to different intervention groups in Stage 2, Stage 2 assignments were not considered in this analysis. Intervention response after Stage 2 was compared based on participants' original Stage 1 group.
Measure: Count of Participants; unit: Participants
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 | Received Low Intensity Frontline Intervention in Stage 1
Number analyzed (Participants) | 328 | 337
Participants
  Week 11-12 | 230 | 198
  Week 24-25 | 194 | 187
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 vs Received Low Intensity Frontline Intervention in Stage 1; Week 12 comparison; Test type: Superiority — Predicted probabilities were estimated using the Stata command "margins" following "melogit," and these probabilities were then expressed as expected percentages; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.28 to 2.64]
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 vs Received Low Intensity Frontline Intervention in Stage 1; Week 25 comparison; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.84 to 1.71]

15. Primary Outcome: Reduction in Methamphetamine Use: Matrix vs. Matrix + CM Adaptive Intervention
Description: Treatment response is defined as testing methamphetamine-negative in 4 out of a possible 4 urine tests during Weeks 24-25.
Time Frame: Week 24-25 (end of stage 2)
Population: Non-responders who were re-randomized to the Matrix intervention in Stage 2 are compared to non-responders who were re-randomized to the Matrix + contingency management in Stage 2; data are aggregated over both Stage 1 interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Received Matrix in Stage 2 | Received Matrix + Contingency Management in Stage 2
Number analyzed (Participants) | 108 | 107
Participants | 13 | 28
Statistical Analysis 1: Comparison: Received Matrix in Stage 2 vs Received Matrix + Contingency Management in Stage 2; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.37 to 6.47]

16. Secondary Outcome: Changes in Quality of Life: High- vs. Low-Intensity Frontline Intervention With Matrix/Matrix + CM in Stage 2
Description: Quality of life will be assessed using the EQ-5D-5L instrument, which includes five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity. Responses will be converted into a single utility index score using the Vietnamese value set (https://doi.org/10.1007/s11136-020-02469-7) ranging from 0-1, where higher scores indicate better health-related quality of life. In addition, participants will rate their overall health on the EQ Visual Analogue Scale (VAS), ranging from 0 ("worst imaginable health") to 100 ("best imaginable health"), with higher scores reflecting better perceived health. Both the EQ-5D-5L utility index and the VAS score will be analyzed as continuous outcomes.
Time Frame: Baseline (start of Stage 1) and week 24 (end of Stage 2)
Population: Only participants classified as Stage 1 non-responders with completed assessments at week 24 were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 | Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 | Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2
Number analyzed (Participants) | 33 | 66 | 41 | 56
score on a scale
  Baseline EQ-5D-5L value | 1.0 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1)
  Baseline VAS | 73.8 (16.4) | 74.4 (15.6) | 73.5 (14.7) | 73.3 (16.0)
  Week 24 EQ-5D-5L value | 1.0 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.2)
  Week 24 VAS | 74.6 (16.4) | 71.4 (17.6) | 72.6 (15.1) | 75.1 (16.9)
Statistical Analysis 1: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Baseline comparison of groups on quality of life value; Test type: Superiority; p = 0.284, Kruskal-Wallis
Statistical Analysis 2: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Baseline comparison of groups on VAS score; Test type: Superiority; p = 0.957, Kruskal-Wallis
Statistical Analysis 3: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison of groups on quality of life value; Test type: Superiority; p = 0.842, Kruskal-Wallis
Statistical Analysis 4: Comparison: Received High Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix in Stage 2 vs Received High Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2 vs Received Low Intensity Frontline Intervention in Stage 1 and Matrix + CM in Stage 2; Week 24 comparison of groups on VAS score; Test type: Superiority; p = 0.611, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period, from June 29, 2021, to April 27, 2024. For each participant, data were collected over a 48-week period, beginning at enrollment and continuing through the 48-week follow-up visit.
Description: Adverse events in this trial are defined as medical issues that do not require hospitalization. Serious adverse events are defined as life-threatening events such (e.g., suicide, opioid overdose) or other events that have a negative impact on participants' life such as incarceration or compulsory drug rehabilitation.
Groups:
- Low Intensity Frontline Intervention: Participants randomized into the low intensity frontline intervention arm (6 weeks of contingency management plus 6 weeks of group education0
- High Intensity Frontline + SMS Reminders: Participants who receive the high intensity frontline intervention and SMS reminders in the adaptive phase
- High Intensity Frontline + Matrix Only: Participants who receive the high intensity frontline intervention and Matrix in the adaptive phase
- High Intensity Frontline + Matrix + Contingency Management: Participants who receive the high intensity frontline intervention and Matrix plus contingency management in the adaptive phase
- Low Intensity Frontline + SMS Reminders: Participants who receive the low intensity frontline intervention and SMS reminders in the adaptive phase
- Low Intensity Frontline + Matrix Only: Participants who receive the low intensity frontline intervention and Matrix in the adaptive phase
- Low Intensity Frontline + Matrix + Contingency Management: Participants who receive the low intensity frontline intervention and Matrix plus contingency management in the adaptive phase
Arm/Group | High Intensity Frontline Intervention | Low Intensity Frontline Intervention | High Intensity Frontline + SMS Reminders | High Intensity Frontline + Matrix Only | High Intensity Frontline + Matrix + Contingency Management | Low Intensity Frontline + SMS Reminders | Low Intensity Frontline + Matrix Only | Low Intensity Frontline + Matrix + Contingency Management
All-Cause Mortality (participants affected / at risk) | 2/328 | 1/337 | 1/230 | 0/40 | 2/45 | 1/198 | 0/68 | 1/62
Serious Adverse Events (participants affected / at risk) | 7/328 | 9/337 | 14/230 | 6/40 | 5/45 | 5/198 | 6/68 | 3/62
Other Adverse Events (participants affected / at risk) | 2/328 | 4/337 | 1/230 | 0/40 | 0/45 | 3/198 | 0/68 | 1/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Intensity Frontline Intervention (N=328) | Low Intensity Frontline Intervention (N=337) | High Intensity Frontline + SMS Reminders (N=230) | High Intensity Frontline + Matrix Only (N=40) | High Intensity Frontline + Matrix + Contingency Management (N=45) | Low Intensity Frontline + SMS Reminders (N=198) | Low Intensity Frontline + Matrix Only (N=68) | Low Intensity Frontline + Matrix + Contingency Management (N=62)
Incarceration (Social circumstances) | 4 (4) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Sent to compulsory drug rehabilitation programs (Social circumstances) | 2 (2) | 2 (2) | 9 (9) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 1 (1) — Participants were sent to compulsory drug rehabilitation programs by the police or by their families.
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Intensity Frontline Intervention (N=328) | Low Intensity Frontline Intervention (N=337) | High Intensity Frontline + SMS Reminders (N=230) | High Intensity Frontline + Matrix Only (N=40) | High Intensity Frontline + Matrix + Contingency Management (N=45) | Low Intensity Frontline + SMS Reminders (N=198) | Low Intensity Frontline + Matrix Only (N=68) | Low Intensity Frontline + Matrix + Contingency Management (N=62)
COVID-19 infection (mild to moderate) (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Accidents and injuries (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Accidents and injuries that do not require hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04706624/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT04706624/ICF_001.pdf